CLINICAL TRIAL: NCT02133664
Title: Lipoic Acid and Omega-3 Fatty Acids for Cognitive Impairment in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Lynne Shinto, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PP2190
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis; Cognition
Keywords: multiple sclerosis; cognition; clinical trial; thiotic acid; Omega-3 fatty acids
MeSH Terms: conditions — Multiple Sclerosis | interventions — Thioctic Acid; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lipoic acid and omega-3 fatty acids (Experimental): lipoic acid and omega-3 fatty acids
  Interventions: Drug: lipoic acid and omega-3 fatty acids
- placebo (Placebo Comparator): placebo oil and placebo lipoic acid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lipoic acid and omega-3 fatty acids — alpha lipoic acid as racemic form at 1,200 mg per day omega-3 fatty acids as fish oil concentrate containing a daily dose of 1.35 grams docosahexanoic acid and 1.95 grams of eicosapentaenoic acid
  Other Names: thiotic acid; fish oil; fish oil concentrate
  Arms: lipoic acid and omega-3 fatty acids
Drug: Placebo — placebo lipoic acid and placebo oil
  Other Names: placebo lipoic acid and placebo oil
  Arms: placebo

SUMMARY:
The primary aim is to collect data to determine the correct effect size on the primary outcome to aid in the design of a larger study: The primary outcome is to determine if lipoic acid and omega-3 fatty acids can improve cognitive function in people with multiple sclerosis that have cognitive dysfunction.

DETAILED DESCRIPTION:
The study is designed as a randomized, double-blind, placebo-controlled pilot trial. The primary aim of the study is to determine if lipoic acid and omega-3 fatty acids can improve cognitive function over 12-weeks in people with multiple sclerosis that have a baseline score of at least two standard deviations below normative values on any one of four cognitive tests that include, Paced Auditory Serial Addition Task (PASAT), Stroop Color-Word Test, California Verbal Learning Test-II (CVLT-II), and Controlled Oral Word Association Test (COWAT).

The secondary aim is to determine treatment effects on markers of endothelial inflammation, insulin dysregulation, and mitochondrial dysfunction that may be related to cognitive dysfunction by measuring soluble intercellular adhesion molecule-1 (sICAM-1) levels, homeostasis model of insulin resistance (HOMA-IR), and MRI phosphorus imaging in a subset of study participants. The study will also measure safety by adverse event reports and laboratory measures; plasma fatty acid levels; serum lipoic acid levels.

ELIGIBILITY:
Inclusion Criteria:

* • A definite diagnosis of multiple sclerosis (MS) with relapsing remitting or secondary progressive course

  * Age 18 to 65 years, inclusive
  * A score two or more standard deviations below the mean in one or more of the following cognitive tests: PASAT, COWAT, CVLT -II, Stroop
  * Expanded Disability Status Scale (EDSS) 0-7.5, inclusive
  * Suboptimal omega-3 levels (plasma docosahexaenoic acid [DHA] + eicosapentaenoic acid [EPA] < 5.0% of total plasma fatty acids)
  * If taking MS disease modifying medications, on stable dose for > 6 months preceding enrollment
  * Able to read and write English

Exclusion Criteria:

* • Moderate to severe depression (Beck Depression Inventory score > 19)

  * Any significant uncontrolled medical problem including diabetes requiring insulin.
  * MS relapse within the 30 days before screening
  * Abnormalities of coagulation or current use of prescription anticoagulants or antiplatelet agents. Aspirin and other nonsteroidal anti-inflammatory drugs (NSAIDs) are not excluded.
  * Fish intake of one 6 ounce serving > once a week less than 2 months prior to enrollment
  * Omega-3 fatty acid supplement intake (e.g. fish oil capsules, cod liver oil) less than 2 months prior to enrollment
  * Lipoic Acid supplementation less than 1 month prior to enrollment
  * Taking systemic corticosteroids, neuroleptics, antiparkinsonian agents, and/or narcotic analgesics. Low dose sinemet and dopamine agonist taken once a day for restless leg syndrome is not an exclusion.
  * Contraindications to MRI, including: subjects with intrathecal pumps, stimulators, pacemakers, aneurysm clips, non-removable hearing aids, or metal fragments in the eyes. Other exclusion criteria include the inability to lie flat on the back for 40 minutes at a time or a self-reported history of claustrophobia. Subjects with a history of hip replacement and those with well-documented, verifiable, MRI-safe cardiac stents will not be excluded from the study.
  * Epilepsy or history of seizures.
  * Pregnancy or women not using a reliable form of contraception
  * Corrected binocular visual acuity worse than 20/50 or more than one error on binocular color vision testing with the Ishihara Color plates or sustained nystagmus or diplopia on primary gaze
  * Inability to complete the neuropsychological test battery at the screening visit
  * Participation in another intervention study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Shinto, ND, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 participants were excluded from the study for the following: did not meet inclusion criteria (i.e. test scores too high, colorblindness, unclear cognitive status), declined to participate, could not consent, lost to follow-up, and started fish oil.
Period: Overall Study
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Started | 26 | 28
Completed | 21 | 21
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Lipoic Acid and Omega-3 Fatty Acids: lipoic acid and omega-3 fatty acids
  Alpha lipoic acid and omega-3 fatty acids: alpha lipoic acid as racemic form at 1,200 mg per day omega-3 fatty acids as fish oil concentrate containing a daily dose of 1.35 grams docosahexanoic acid and 1.95 grams of eicosapentaenoic acid
- Total: Total of all reporting groups
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 28 | 53
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.34 (10.91) | 52.96 (8.85) | 51.22 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Paced Auditory Serial Addition Task (PASAT)
Description: The PASAT is a measure of working memory and sustained attention frequently used in multiple sclerosis treatment outcome studies. The examinee is presented with a series of numbers at 2 second intervals on an audiotape and responds by always adding the last two numbers on the tape before the next number is presented. The change in total number of correct responses from baseline to 12 weeks is the measurement for the outcome.
Time Frame: Baseline to 12 weeks
Population: Only participants who completed PASAT at both baseline and 12 weeks were analyzed.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 21 | 21
correct responses | 2.24 (4.69) | 3.38 (5.46)
Statistical Analysis 1: Comparison: Lipoic Acid and Omega-3 Fatty Acids vs Placebo; With the initial sample size plan of 53 subjects, we expect an 80% power to detect a significant difference in PASAT score with a mean difference of 8.3 points between the treatment and placebo group; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-2.03 to 4.32], Standard Error of Mean 1.57

2. Primary Outcome: Stroop Color-Word Test
Description: The Stroop test assess attention and executive function.The task consists of 3 tasks with only red, green, and blue colors used. The first task asks the subject to name the colors of spots on cards. If a subject can perform this task the second task is performed in which a subject must read the names of colors listed on cards (which are printed in congruent colors). In the third task, the subject is shown a series of words naming colors but the words and colors are mismatched; so the word "yellow" may be red, the word "blue" may be green and so forth. The subject is instructed to ignore the word and name the color. The subject will have the tendency to read the word rather than name the color, the so-called Stroop effect. This third part of the test is referred to as the interference condition and is the critical measurement. The change in time it takes to complete the interference from baseline to 12 weeks is the outcome measure.
Time Frame: baseline to 12 weeks
Population: Analysis occurs only for participants who completed Stroop at both baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 23 | 23
seconds | -5.59 (12.77) | -2.87 (7.01)

3. Primary Outcome: California Verbal Learning Test-II (CVLT-II)
Description: CVLT-II is a measure of verbal learning/memory. It is comprised of lists containing 16 words, each of which fit into one of four categories of "shopping list" items. Five trials are administered followed by presentation of a different list. Free and cued recall of the original list is assessed. The change in long delay free recall from baseline to 12 weeks will be the measurement used for outcome.
Time Frame: baseline to 12 weeks
Population: Only participants who completed CVLT-II at baseline and 12 weeks were analyzed
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 23 | 23
correct responses | 1.57 (1.85) | 1.65 (2.44)

4. Primary Outcome: Controlled Oral Word Association Test (COWAT)
Description: The COWAT is a letter fluency test. Participants are asked to generate as many words as possible beginning with a particular letter of the alphabet during one minute. Alternate versions using 3 letters are used for each examination. The change in total number of words produced for the 3 letters from baseline to 12 weeks will be the outcome.
Time Frame: baseline to 12 weeks
Population: Only participant who completed COWAT at both baseline and 12 weeks were analyzed
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 23 | 23
words | 0.70 (7.71) | 0.39 (7.14)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/28
Other Adverse Events (participants affected / at risk) | 21/26 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lipoic Acid and Omega-3 Fatty Acids (N=26) | Placebo (N=28)
Kidney Infection (Renal and urinary disorders) | 1 | 0 — Hospitalized 7/6/15-7/10/15 and treated for kidney infection and dehydration.
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 — Participant went on an airplane- during descent, lost hearing in right ear.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lipoic Acid and Omega-3 Fatty Acids (N=26) | Placebo (N=28)
Throat irritation (Gastrointestinal disorders) | 3 | 0 — Burning in throat
Dysphagia (Gastrointestinal disorders) | 0 | 2 — Difficulty swallowing study supplement
Fall (Injury, poisoning and procedural complications) | 0 | 4
Fatigue (General disorders) | 3 | 1
Adverse drug reaction (Gastrointestinal disorders) | 2 | 0 — Fishy taste, fish burps
Headache (Nervous system disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1 — Indigestion
Nausea (Gastrointestinal disorders) | 6 | 2
Urine odor abnormal (Renal and urinary disorders) | 4 | 0 — Strong odor to urine
Incontinence (Renal and urinary disorders) | 2 | 1
Urinary tract infection (Renal and urinary disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes